CLINICAL TRIAL: NCT06393556
Title: Assessment and Minimization of Preoperative Fear of the Unknown Using a VR Experience of the Theatre Suite; a Randomized Control Trial
Brief Title: VR for the Reduction of Perioperative Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Gold Coast Hospital and Health Service (Other Government)
Responsible Party: Principal Investigator, Günther Rezniczek, Head of Ob/Gyn Research Lab (MHH), Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: VRPERIOP1
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Anxiety State
Keywords: anxiety; virtual reality; gynecologic-oncological surgery
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care provider measuring the primary outcome scale at T2 was not aware of the intervention given at T0/1. Statistical data analysis initially was prepared not knowing which group was the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): Care-as-usual + virtual reality intervention during a pre-operative visit
  Interventions: Other: Virtual reality experience
- Control (No Intervention): Care-as-usual during a pre-operative visit

INTERVENTIONS:
Other: Virtual reality experience — An immersive VR experience, delivered using a VR head-mounted display, of the real-world environment at the hospital, featuring the pre-operative admission suite, pre-anesthetic bay, operating theatre, postoperative recovery room, and medical staff.
  Arms: Virtual reality

SUMMARY:
The study, set to take place at Gold Coast University Hospital in Australia, will be conducted as a randomized controlled trial. Patients preparing for gynecological cancer surgery will be recruited and randomly assigned to one of two groups: those who will receive standard care plus a virtual reality (VR) intervention, and those who will receive only standard care. Standard care encompasses the usual pre-operative procedures and support provided by the hospital staff.

We hypothesize that immersing patients in a preparatory virtual environment that shows them what they are to expect during their upcoming hospital stay for surgery, could help reduce their anxiety levels.

DETAILED DESCRIPTION:
The study objective is to determine whether exposure to the operating theatre suite via virtual reality (VR) for patients undergoing gynecologic-oncological surgery reduces pre-operative anxiety.

After patients are recruited, their anxiety level is measured by a simple 6-item visual anxiety scale (T0). Patients are then randomized into either receiving care-as-usual (CAU), or CAU combined with a VR experience (~3.5 minutes; with background music and narration) where they are familiarized with the environment they will encounter during their stay for their cancer operation. Anxiety is measured again (T1). Days/weeks later, when patients are back in the hospital for their surgery (T2), anxiety is measured again in the preanesthetic bay, before receiving any anesthetics. Personnel collecting the anxiety scale at T2 will be unaware whether a patient had received the VR intervention or not.

Randomization will be performed by a person unrelated to the study by using a computerized randomization tool to generate an allocation list and inserting paper slips with the group allocation into consecutively numbered, opaque envelopes which are opened, in order, at the time of randomization.

Using a two-sided Wilcoxon-Mann-Whitney test and targeting a power of 80% at a significance level α of 0.05, abd assuming a clinically relevant difference in the anxiety scale of at least one "face" (i.e. at least 1 point on the 6-item scale) between the two groups and a within-group standard deviation of 1.6 (effect size: 0.625), sample size was determined as 34 patients per group for a 1:1 group allocation. Assuming a drop out/lost-to-follow up rate of up to 15%, 80 patients (40 per group) are to be recruited.

Descriptive statistic analysis will be performed. Within-group and between-group assessements will be done using Wilcoxon signed rank test and the Mann-Whitney rank sum test, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Gynecological oncology patients with scheduled surgery

Exclusion Criteria:

* Language barrier
* Inability to provide consent
* Having undergone any procedure at the operating theatre in the previous 5 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Anxiety | T0 (before randomization), T1 (same day as T0, but after care as usual +/- VR; usually inside 1 hour), T2 (days/weeks later, before surgical procedure - exact gap is unknown; expected: >3 days, median around 4-7 weeks)
  Anxiety level measured by a 6-item visual scale (1 .. least anxiety, 6 ... highest anxiety)

CONTACTS AND LOCATIONS:
Overall Officials: Bernd C Schmid, MD, Principal Investigator — Gold Coast University Hospital
Locations (1):
- Gold Coast University Hospital, Southport, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared upon reasonable request for purposes that have been approved by the respective Institutional Review Board
Supporting Information: Study Protocol, ICF
Time Frame: After publication
Access Criteria: Reasonable request; approval of intended use by an Institutional Review Board

REFERENCES:
- [Background] Cao X, Yumul R, Elvir Lazo OL, Friedman J, Durra O, Zhang X, White PF. A novel visual facial anxiety scale for assessing preoperative anxiety. PLoS One. 2017 Feb 14;12(2):e0171233. doi: 10.1371/journal.pone.0171233. eCollection 2017. PMID 28196099
- [Result] Schmid BC, Marsland D, Jacobs E, Rezniczek GA. A Preparatory Virtual Reality Experience Reduces Anxiety before Surgery in Gynecologic Oncology Patients: A Randomized Controlled Trial. Cancers (Basel). 2024 May 17;16(10):1913. doi: 10.3390/cancers16101913. PMID 38791991